CLINICAL TRIAL: NCT02797041
Title: REal Life, Retrospective Study of BOrtezomib Use as secoND Treatment for Myeloma Patients Previously Exposed to Bortezomib-based Therapies as First Line
Brief Title: Bortezomib as First Salvage Therapy for Myeloma Patients Previously Exposed to Bortezomib as Initial Treatment.
Acronym: REBOUND
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: IRCCS Centro di Riferimento Oncologico della Basilicata (Other)
Responsible Party: Principal Investigator, Pellegrino Musto, Scientific Director, IRCCS Centro di Riferimento Oncologico della Basilicata
Other Study IDs: CentroROB
Record Dates: First submitted 2016-06-02; First posted 2016-06-13 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Bortezomib; Relapsed multiple myeloma; Rechallenge
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bortezomib — Re-challenge with bortezomib as second line therapy in myeloma patients relapsed after a previous bortezomib-based treatment
  Other Names: No other drugs evaluated

SUMMARY:
This observational, non-interventional, retrospective, multicenter, national study focuses on collecting information about the effectiveness and safety of bortezomib re-use at first relapse in MM patients already treated in their first line with a bortezomib-based regimen, re-challenged with the same drug according to current clinical practice and/or Italian SIE/SIES/GITMO, IMWG and/or NCCN Guidelines/Treatment Recommendations.

Data will be collected retrospectively from approximately 25 haematologic/oncologic sites in Italy. Approximately, data of up to 100 patients will be collected.

ELIGIBILITY:
Inclusion Criteria:

Patients satisfying all of the following criteria will be enclosed in the study:

* Age ≥ 18 years old
* Patients with documented multiple myeloma that received bortezomib-based regimens as first line treatment (both in clinical practice or clinical trials) even if followed by ASCT (Autologous stem cell transplantation) and that after their first line treatment's clinical or biochemical relapse received again a bortezomib-based treatment according to current clinical practice and/or Italian Societies of Hematology (SIE), Experimental Hematology (SIES) and Transplantation (GITMO), International Myeloma Working group (IMWG) and/or National Cancer Comprehensive Cancer Network (NCCN) guidelines/treatment recommendations.
* Signed Informed Consent form if feasible

Exclusion Criteria:

* Patients not treated with bortezomib as first line therapy and/or second line therapy
* Patients with more than one relapse before bortezomib re-use
* Patients unable to understand and sign Informed Consent form (see exceptions listed in section 8 "Informed consent")
* Patients who received bortezomib at relapse in combination with any investigational drug not-approved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with documented multiple myeloma that received bortezomib-based regimens as first line treatment and that after their first line treatment's relapse received again a bortezomib-based treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Response rate | March, 31, 2016
  International Myeloma Study Group Criteria
Adverse events | March,31, 2016
  Types (haematological and non hematological) and degree (Common terminology criteria adverse criteria)

SECONDARY OUTCOMES:
Progression free survival 1 and 2 | March, 31, 2016
Time to next treatment | March, 31, 2016
Overall survival | March, 31, 2016
Secondary primary malignancies | March, 31, 2016
  Types and incidence

CONTACTS AND LOCATIONS:
Overall Officials: Pellegrino Musto, MD, Principal Investigator — IRCCS Centro di Riferimento Oncologico della Basilicata, Rionero in Vulture (Pz), Italy

IPD SHARING:
Plan to Share IPD: Yes
Central database of single patients